CLINICAL TRIAL: NCT06413264
Title: Ultrasonography Guided Pneumoperitoneum for Laparoscopic Surgery in Morbidly Obese Patients: A Single-blinded Randomized Control Study (USP TRIAL)
Brief Title: Ultrasonography Guided Pneumoperitoneum for Laparoscopic Surgery in Morbidly Obese Patients
Acronym: USP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Dr. Prakash Kumar Sasmal, Professor of General Surgery, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: T/IM-NF/Gen.Surg/23/118
Record Dates: First submitted 2024-04-28; First posted 2024-05-14 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Pneumoperitoneum; Morbid Obesity; Bariatric Surgery Candidate
Keywords: pneumoperitoneum; closed technique; Veress needle; ultrasonography-guided; morbidly obese; bariatric surgery; metabolic surgery; access-related injury
MeSH Terms: conditions — Pneumoperitoneum; Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: Single blinded randomised controlled study where only the patient is blinded
Who Masked: Participant
Masking Description: Only patients will be blinded about the allocations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- USG-guided Veress needle insertion (Experimental): Ultrasonography-guided Veress needle will be inserted, and a real-time pneumoperitoneum will be created as the first step of a laparoscopic bariatric surgical procedure. The bariatric procedures include laparoscopic sleeve gastrectomy and gastric bypass procedures. The ultrasound's high-frequency (10-13Hz) linear probe will be used peri-operatively to identify the planes of the abdominal wall. Once the Veress needle is successfully inserted into the peritoneal cavity in real-time visualisation and pneumoperitoneum created, thereafter the bariatric procedures will be continued as routinely done.
  Interventions: Procedure: Ultrasonography guided Veress needle insertion for creating pneumoperitoneum
- Blind Veress needle insertion (Active Comparator): The Veress needle is inserted blindly, as regularly done in any other laparoscopic surgery, and the successful pneumoperitoneum is confirmed by aspiration of the needle, saline drop test and percussion on the abdomen.
  Interventions: Procedure: Veress needle will be inserted blindly as a closed technique for creating pneumoperitoneum

INTERVENTIONS:
Procedure: Ultrasonography guided Veress needle insertion for creating pneumoperitoneum — A real-time visualisation of the path of the Veress needle entry by the use of high frequency (13-6 MHz) probe ultrasonography.
  Other Names: Sonosite Edge II Portable Ultrasound machine
  Arms: USG-guided Veress needle insertion
Procedure: Veress needle will be inserted blindly as a closed technique for creating pneumoperitoneum — The Veress needle is inserted blindly and guided by the resistance of tissues and the click sounds of layers of abdominal wall.
  Other Names: Stainless steel spring loaded reusable hollow needle of 2mm in diameter and 15-18cm long
  Arms: Blind Veress needle insertion

SUMMARY:
Bariatric Surgery for morbid obesity is indicated when BMI > 40 kg/m2 without comorbidities or BMI > 35 kg/m2 with co-morbidities. Different surgeries performed for obesity are classified as restrictive, malabsorptive, and hybrid procedures.

Because laparoscopic surgery has increased the interest and growth of bariatric surgery, soaring demand for laparoscopic bariatric surgery from patients has boosted the boom in bariatric surgery worldwide.

Achieving pneumoperitoneum is the initial and one of the most crucial steps in any laparoscopic surgery, giving the surgeon working space to operate on a particular organ/organ system. Usually, pneumoperitoneum is achieved either by a closed technique with a veress needle or an open technique with many variations like finger assisted or the conventional open technique.

Given the excess amount of subcutaneous fat in morbidly obese patients, putting a veress needle to achieve pneumoperitoneum successfully is particularly challenging which takes a toll on the operating surgeon when he/she is trying to locate the midline one can either overshoot to cause omental emphysema or undershoot getting lost in the subcutaneous fat. It is usually done in the supra umbilical area. Sometimes, due to previous surgical scars other sites are preferred.

Sonography is routinely used by radiologists with negligible radiation exposure. Anesthesiologists in the operating room have used it for many assisted procedures like central line insertion / giving nerve blocks. It can also be used in obese patients undergoing metabolic surgery to assist in creating pneumoperitoneum by a veress needle.

Advantages of Intraoperative ultrasonography in this particular study :

1. To quantify the thickness of subcutaneous fat
2. To visualise the linea alba and guide the veress needle safely into the peritoneal cavity
3. Real-time visualisation of the pneumoperitoneum created
4. Avoid complications like omental emphysema, bowel or vascular injury

DETAILED DESCRIPTION:
All patients above the age of 18 years with morbid obesity planned for Laparoscopic bariatric surgery will be considered for inclusion in the study. The patient will be explained about the study and asked to sign an informed consent form. The patient's eligibility for the study will be checked by a competent radiologist through pre-operative ultrasonography. All patients will undergo metabolic surgery by a single competent surgeon per the standard operating protocol under general anaesthesia. A single dose of prophylactic antibiotic will be administered 30 minutes before the incision, the patient will be well strapped, and the port sites will be measured and marked. In group A, Ultrasonography will be used to locate the midline precisely and for subsequent puncturing with a Veress needle to enter the peritoneal cavity and the pneumoperitoneum created under real-time vision. In group B, the veress needle is inserted blindly, as regularly done in any other laparoscopic surgery, and the successful pneumoperitoneum is confirmed by percussion on the abdomen. Time taken and the number of attempts for achieving pneumoperitoneum and complications, if any, in both groups will be recorded by an independent assessor.

Sample size calculation :

There are no similar studies done before to assess the role of Ultrasonography in achieving pneumoperitoneum. Hence, the sample size was calculated for a pilot study, as per the recommendation of Sim J and Lewis M, considering precision, proportion, and efficiency. The trial was planned through a study of a continuous variable in two independent, Blind vs. USG guided Veress needle insertions to determine if the two study groups differ in the time taken to start pneumoperitoneum successfully.

The study used for calculating sample size :

Total sample size: 20 in each arm Blinding: Single blinded where only the patient is blinded

ELIGIBILITY:
Inclusion Criteria:

* All patients in the age group of 18 -65 years undergoing laparoscopic bariatric surgery with weight >100 kg
* Subcutaneous fat thickness of more than 5 cm as determined by pre-operative ultrasonography
* BMI > 40 kg/m2

Exclusion Criteria:

* Patients who don't give consent and do not understand the nature of the study
* Patients undergoing a re-do surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Time taken to successfully insert the Veress needle (supra umbilical) into the peritoneal cavity in both arms. | Time taken till the Veress needle tip enters the peritoneal cavity (Maximum allowed time up to 2 minutes). Beyond the time, the Veress needle to be attempted insertion at other sites, including the Palmer's point.
  The time in seconds between the first attempt to insert the Veress needle into the peritoneal cavity and the onset of successful pneumoperitoneum (confirmed by either ultrasonography/saline drop/percussion) in morbidly obese patients undergoing laparoscopic bariatric procedures. A comparison of the time taken to successfully place the Veress needle in the peritoneal cavity by ultrasonography-guided insertion and by blind technique will be made.

SECONDARY OUTCOMES:
Number of attempts to successful Veress needle insertion | Veress needle tip enters the peritoneal cavity (Upto maximum 3 attempts within 2 minutes). Beyond the number of attempts or time, the Veress needle to be attempted insertion at other sites, including the Palmer's point.
  The number of attempts of Veress needle insertion made before successful intraperitoneal placement (confirmed by either ultrasonography/saline drop/percussion) in morbidly obese patients undergoing laparoscopic bariatric procedures. A comparison of the number of attempts of Veress needle insertion to successfully place it in the peritoneal cavity by ultrasonography-guided insertion and by the blind technique will be made.
Incidences of complications out of Veress needle insertion for creating pneumoperitoneum | At the beginning of the laparoscopic surgical procedure, during the diagnostic laparoscopy, the complications (omental emphysema, bowel /vascular injury), if any inadvertently done will be recorded
  To compare the incidence of complications like omental emphysema, bowel injury and vascular injury.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Prakash K. Sasmal, MS, FACS, Principal Investigator — Professor of General Surgery, All India Institute of Medical Sciences, Bhubaneswar, India
Locations (1):
- All India Institute of Medical Sciences, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No
The study outcome will be shared after the end of the trial. An interim study outcome will be shared after half of the study subjects are recruited.